CLINICAL TRIAL: NCT02861235
Title: Comparison Between Myocardial Tomoscintigraphies Using a Semiconductor Camera or a Conventional Camera According to Conditions of Examination Execution: Assessment of Infarction or Ischemia, Injected Dye and Sequence of Injections
Brief Title: Comparison Between Myocardial Tomoscintigraphies Using a Semiconductor Camera or a Conventional Camera
Acronym: DSPECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2009-A00422-55
Record Dates: First submitted 2016-07-29; First posted 2016-08-10 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Myocardial Infarction; Ischemia
MeSH Terms: conditions — Myocardial Infarction; Ischemia | interventions — Gamma Cameras

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1. stress thallium-201 tomoscintigraphy (Experimental)
  Interventions: Other: Stress thallium-201 tomoscintigraphy, followed by a second rest tomoscintigraphy if necessary
- 2. stress technetium-99m tomoscintigraphy 1 (Experimental)
  Interventions: Other: Rest technetium-99m tomoscintigraphy followed by stress technetium-99m tomoscintigraphy on the same day
- 3. stress technetium-99m tomoscintigraphy 2 (Experimental)
  Interventions: Other: Stress technetium-99m tomoscintigraphy followed by rest technetium-99m tomoscintigraphy on the same day
- 4. stress technetium-99m tomoscintigraphy 3 (Experimental)
  Interventions: Other: stress technetium-99m tomoscintigraphy followed by rest technetium-99m tomoscintigraphy in two different days
- 5. rest thallium-201 tomoscintigraphy (Experimental)
  Interventions: Other: Rest thallium-201 tomoscintigraphy with gamma-camera and D.SPECT camera
- 6. rest technetium-99m tomoscintigraphy (Experimental)
  Interventions: Other: Rest technetium-99m tomoscintigraphy with gamma-camera and D.SPECT camera

INTERVENTIONS:
Other: Stress thallium-201 tomoscintigraphy, followed by a second rest tomoscintigraphy if necessary — with gamma-camera and D.SPECT camera
  Arms: 1. stress thallium-201 tomoscintigraphy
Other: Rest technetium-99m tomoscintigraphy followed by stress technetium-99m tomoscintigraphy on the same day — with gamma-camera and D.SPECT camera, in Toulouse centre
  Arms: 2. stress technetium-99m tomoscintigraphy 1
Other: Stress technetium-99m tomoscintigraphy followed by rest technetium-99m tomoscintigraphy on the same day — with gamma-camera and D.SPECT camera, in Nancy centre
  Arms: 3. stress technetium-99m tomoscintigraphy 2
Other: stress technetium-99m tomoscintigraphy followed by rest technetium-99m tomoscintigraphy in two different days — with gamma-camera and D.SPECT camera, in Paris centre
  Arms: 4. stress technetium-99m tomoscintigraphy 3
Other: Rest thallium-201 tomoscintigraphy with gamma-camera and D.SPECT camera — rest thallium-201 tomoscintigraphy for myocardial viability assessment
  Arms: 5. rest thallium-201 tomoscintigraphy
Other: Rest technetium-99m tomoscintigraphy with gamma-camera and D.SPECT camera — rest technetium-99m tomoscintigraphy for myocardial viability assessment
  Arms: 6. rest technetium-99m tomoscintigraphy

SUMMARY:
Myocardial perfusion tomoscintigraphy is a routine medicine procedure to check for the presence and severity of abnormalities of myocardial perfusion, as well as the extension of infarction residua. However, actual imagery devices (gamma cameras) have low resolution and detection sensitivity. A new semiconductor camera has 8 to 10 time higher detection sensitivity and could allow proportionally diminishing injected activities or recording times. Only one pilot study has been recently published on this type of camera, the D.SPECT camera.

This study will compare images recorded during 15 to 20 minutes by conventional cameras and 2 to 4 minutes by D.SPECT camera in patients doing tomoscintigraphy under usual conditions. The purpose is to demonstrate the equivalence of images recorded by two camera types for diagnostic information and the secondary purpose is to demonstrate the superiority of the D.SPECT camera in terms of image quality.

DETAILED DESCRIPTION:
This study will be conducted in Nuclear Medicine departments (Nancy Hospital, Bichat Hospital in Paris, Pasteur private hospital in Toulouse), with D.SPECT camera (Cyclopharma). The D.SPECT camera recording will be realized following the conventional camera recording and will not modify the routine programmed examination. Recording times of D.SPECT camera will be maximum 2 minutes for imaging with a strong activity of technetium-99m labeled dye and maximum 4 minutes for imaging with thallium-201 or with a low activity of technetium-99m labeled dye.6 study groups will be analyzed: 4 groups of patients initially doing stress tomoscintigraphy with thallium-201 (group 1) or with technetium-99m labeled dye and then testing 3 principal injection sequences (group 2, 3, 4), and 2 groups of patients initially doing "myocardial viability" assessment with rest tomoscintigraphy with thallium-201 (group 5) or technetium-99m labeled dye.

Recording comparison obtained with 2 cameras will be done according to qualitative and quantitative criteria on image quality and analyzing diagnosis concordance (presence, type and severity of observed abnormalities).

ELIGIBILITY:
Inclusion Criteria:

* Understanding and signature of informed consent
* Without any contraindication for tomoscintigraphy and stress techniques according to French Society of Cardiology and Nuclear Medicine criteria, as established for all patients doing this routine examination
* Not in emergency situation and with a stable clinical status (without any sign of heart or coronary failure, without uncontrolled high blood pressure under treatment)
* Having an effective contraception for women of childbearing potential

Exclusion Criteria:

* Patient under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2009-11; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Ejection fraction of link ventricle | day 0
Telesystolic volume of link ventricle | day 0
Telediastolic volume of link ventricle | day 0
Diagnosis of stress ischemia with Myocardial Tomoscintigraphy data | day 0
Area of damaged regions of heart | day 0

SECONDARY OUTCOMES:
Global myocardial activity | day 0
Qualitative score of image quality | day 0

CONTACTS AND LOCATIONS:
Overall Officials: Wassilia DJABALLAH, Principal Investigator — Service de Médecine Nucléaire, Hôpital de Brabois, 54500, Vandoeuvre-les-Nancy, France
Locations (3):
- France (3):
  - Service de Médecine Nucléaire, Hôpital de Bichat, Assistance Publique des Hôpitaux de Paris, Paris
  - Service de Médecine Nucléaire, Clinique Louis Pasteur, Toulouse
  - Service de Médecine Nucléaire, Hôpital de Brabois, CHU de Nancy, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No